CLINICAL TRIAL: NCT04563858
Title: Interdisciplinary Treatment Towards a Patient With Delirium
Brief Title: Polish Validation 4AT Tool
Status: Completed | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Collaborators: University of Rzeszow (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lucyna Tomaszek, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: 9/05/2020
Record Dates: First submitted 2020-09-19; First posted 2020-09-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Delirium, Postoperative; Surgical Procedure
Keywords: Delirium; 4AT Scale; Cardiac surgery; Validation
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac patients
  Interventions: Diagnostic Test: Validation

INTERVENTIONS:
Diagnostic Test: Validation — Assessment of Polish version of the 4AT

SUMMARY:
Delirium is a phenomenon which affects patients with various disorders and representing various age groups. Screening instruments make it possible to diagnose the condition at an early stage and to prevent its development. The aim of the study is to examine the reliability and validity of the Polish version of the 4AT (Pol4-AT) in patients after cardiac surgery.

Procedure of validation:

After obtaining the author's consent, the original English version of the 4AT was separately translated by 3 centres working on the validation of the Pol4-AT (University of Rzeszów, Poland; University Hospital in England; Karolinska University, Sweden). Then, three translations were compared, to be approved by the project supervisor (Karolinska University). Any doubts arising during the comparison were consulted with the English translator. As a result, one coherent version was accepted and translated back into English. The questionnaire was distributed in a convenient sample of 20 patients to examine the validity of the face. Vague words and statements were changed, and the final version translated into Polish was created. The Pol4-AT was tested for internal consistency and reliability.

DETAILED DESCRIPTION:
Delirium, which generally is triggered by underlying medical conditions, is an acute and fluctuating disorder associated with attention and cognitive defects, and frequently accompanied by excessive arousal and perception-related problems. Delirium may lead to a variety of complications, e.g. cognitive impairments. Development of delirium is promoted by both anaesthesia and pain. Patients subjected to cardiac surgeries are at risk of delirium due to such factors as extracorporeal circulation applied during the intervention and various cardiovascular complications. Rapid identification of the problem may help eliminate avoidable complications which can be prevented at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* adults
* able to sign the consent form
* elective cardiac surgery
* extracorporeal circulation

Exclusion Criteria:

* unconscious patients
* diagnosed mental illness
* patient's lack of consent to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Validity for the Polish version 4AT | third day following a surgery
  The Pol4-AT questionnaire consists of 4 items assessing four aspects of delirium: alertness, short mental test, attention, acute change or fluctuating course.
  A 4AT total score of 0 indicates that delirium or cognitive impairment is unlikely; a score between 1 and 3 indicates possible cognitive impairment and a score ≥ 4 is suggestive of delirium.
Reliability for the Polish version 4AT | third day following a surgery
  The Pol4-AT questionnaire consists of 4 items assessing four aspects of delirium: alertness, short mental test, attention, acute change or fluctuating course.
  A 4AT total score of 0 indicates that delirium or cognitive impairment is unlikely; a score between 1 and 3 indicates possible cognitive impairment and a score ≥ 4 is suggestive of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Krupa, PhD, Study Director — Medical College of Rzeszow University Institute of Health Sciences
Locations (1):
- Medical College of Rzeszow University Institute of Health Sciences, Rzeszów, Warzywna Saint 1, Poland